CLINICAL TRIAL: NCT05154799
Title: Developmental Coordination Disorder: Role of Perceptual Deficits and Body Representation
Brief Title: Developmental Coordination Disorder
Acronym: DYSENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL21_0338
Record Dates: First submitted 2021-07-08; First posted 2021-12-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Motor Skills Disorders; Neurodevelopmental Disorders
Keywords: Healthy subject; Developmental coordination disorder
MeSH Terms: conditions — Motor Skills Disorders; Neurodevelopmental Disorders | interventions — Proprioception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dyspraxic children (Experimental): Children with Developmental coordination disorder
  Interventions: Behavioral: Proprioception and tactile localization with manual or ocular response and/or free hand grasp
- Control children (Experimental): Healthy children
  Interventions: Behavioral: Proprioception and tactile localization with manual or ocular response and/or free hand grasp
- Dyspraxic adults (Experimental): Adults with with Developmental coordination disorder
  Interventions: Behavioral: Proprioception and tactile localization with manual or ocular response and/or free hand grasp
- Control adults (Experimental): Control adults
  Interventions: Behavioral: Proprioception and tactile localization with manual or ocular response and/or free hand grasp

INTERVENTIONS:
Behavioral: Proprioception and tactile localization with manual or ocular response and/or free hand grasp — In the first part of the study, the subject must designate a target in 2 ways: manual pointing or ocular saccadic response.
  In the second part of the study the subject will have to reach and grasp a rectangular block of wood placed on the table at a distance of 35 cm. He will have to catch the wooden block, lift it a few centimeters and put it back on the table. Tool use and control phases: the subject grasps the wooden block with a tool or without the tool but with a weighted bracelet loading his wrist by the same amount as the tool.

SUMMARY:
Developmental Coordination Disorder (DCD) corresponds to a clumsiness, a slowness and an inaccuracy of motor performance. This neurodevelopmental disorder affects 6% of school-aged children, and disturbs daily life activities and academic performances. The etiology of DCD is still unknown. An understanding of this disorder is necessary to improve interventions and therefore quality of life of these people.

A deficit of the so-called internal models is the most commonly described hypothesis of DCD. Indeed, children with DCD exhibit difficulties in predictive control. Internal models, useful for motor control, are closely related to the sensory system, as they are elaborated on and constantly fed by sensory feedback. Deficits in sensory performance are described in DCD, mostly in the visual system, which could in turn partly explain poor motor performance. However, visuo-perceptual deficits cannot explain the entire motor difficulties because some activities in daily life, as buttoning a shirt, are often performed without visual control. Although the integrity of proprioceptive and tactile systems is necessary for the building of internal models, and therefore for a stable motor control, these sensory systems have been very little investigated in DCD.

Moreover, using a tool is often disturbed in children with DCD. In neurotypical subjects, tool use induces a plasticity of body representation, as reflected by modifications of movement kinematics after tool use. Proprioceptive abilities are necessary for this update of the body schema. Thus, potential deficits of the proprioceptive system in children with DCD could impair the plastic modification of the body schema, and hence of motor performance, when using a tool. The aim of this study is to identify the main cause of the DCD, both by evaluating the tactile and proprioceptive abilities and by assessing the body schema updating abilities in children with DCD.

While some daily life activities improve with age, some motor difficulties persist in adults with DCD. To our knowledge, perceptual abilities have never been investigated in adults with DCD and it is thus unknown whether perceptual deficits are still present in adulthood. This information could allow us to understand if motor difficulties in adult DCD are caused by enduring perceptual deficits and/or impaired plasticity of body schema. The second aim of this study is to evaluate abilities of perception and of body schema plasticity in adults with DCD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 9 to 11 or 18 to 40
* Affiliated to a health care organism
* Signed written informed consent (adult subjects)
* One of the legal guardians of children subjects providing their free, informed and written consent to participate in the study; With the child also giving orally his consent to participate.

For participants with Developmental coordination disorder:

* Subjects fulfilling the diagnostic criteria for dyspraxia of DSM-5 (these criteria will be verified by the principal investigator)
* Total MABC-2 score below the 15th percentile (if this MABC-2 assessment is already available).

Exclusion Criteria:

* Prematurity
* Known neurological pathology (other than dyspraxia)
* Intellectual disability
* Visual impairment
* Surgery or trauma to the upper limbs that has occurred too recently to allow proper testing
* Subject under tutorship or curatorship
* Subject deprived of liberty by a judicial or administrative decision

For healthy volunteers only:

- History of developmental coordination disorder in close relatives (parents, children, siblings).

Ages: 9 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2027-01-21 (Estimated); Study Completion 2027-01-21 (Estimated)

PRIMARY OUTCOMES:
Localization error distance | At day 1
  Difference in localization error distance between manual response and ocular response: measure in mm between the target and the response of the subject.
  Task 1 : proprioceptive localization with manual response Task 2 : proprioceptive localization with ocular response Task 3: tactile localization with manual response Task 4: tactile localization with ocular response
  In the 4 tests, we will measure the deviation (in mm) between the localization response of the subject and the reference point.
  For tasks 1 and 2, the reference point is the position of the hidden index finger of the subject.
  For tasks 3 and 4, the reference point is the position of the tactile stimulation applied to the hidden arm of the subject.
  For the manual response, the subject must designate with his other index finger where he considers the target to be.
  For the ocular saccadic response, the subject must shift his gaze and look where he considers the target to be.

SECONDARY OUTCOMES:
Reaction time of motor localization response | At day 1
  A difference between 'go signal' and initiation of localization motor responses (Tasks 1-4) measured in msec
change related to tool-use of amplitude of velocity peak and the peak opening of the thumb-index grip of free reach-to-grasp limb movements | At day 1
  the subject will perform free reach-to-grasp limb movements before and after a tool-use phase (grasping a wooden block with a mechanical clamp) or a control phase (grasping the block without tool but with a bracelet loading the wrist by the same amount as the tool). For both tool-use and control conditions, the pre- versus post- difference of trajectory of free reach-to-grasp limb movements will be computed with amplitude in mm/sec of velocity peak and the peak opening of the thumb-index grip.
change related to tool-use of latency of velocity peak and the peak opening of the thumb-index grip of free reach-to-grasp limb movements | At day 1
  the subject will perform free reach-to-grasp limb movements before and after a tool-use phase (grasping a wooden block with a mechanical clamp) or a control phase (grasping the block without tool but with a bracelet loading the wrist by the same amount as the tool). For both tool-use and control conditions, the pre- versus post- difference of trajectory of free reach-to-grasp limb movements will be computed with latency in msec of velocity peak and the peak opening of the thumb-index grip.
change related to tool-use of acceleration peak of the upper limb of free reach-to-grasp limb movements | At day 1
  the subject will perform free reach-to-grasp limb movements before and after a tool-use phase (grasping a wooden block with a mechanical clamp) or a control phase (grasping the block without tool but with a bracelet loading the wrist by the same amount as the tool). For both tool-use and control conditions, the pre- versus post- difference of trajectory of free reach-to-grasp limb movements will be computed with acceleration peak in mm/sec2 of the upper limb.
change related to tool-use of deceleration peak of the upper limb of free reach-to-grasp limb movements | At day 1
  the subject will perform free reach-to-grasp limb movements before and after a tool-use phase (grasping a wooden block with a mechanical clamp) or a control phase (grasping the block without tool but with a bracelet loading the wrist by the same amount as the tool). For both tool-use and control conditions, the pre- versus post- difference of trajectory of free reach-to-grasp limb movements will be computed with deceleration peak in mm/sec2 of the upper limb.

CONTACTS AND LOCATIONS:
Overall Officials: Denis PELISSON, Dr, Principal Investigator — Centre de Recherche en Neurosciences de Lyon
Locations (1):
- Equipe IMPACT du CRNL INSERM U1028, CNRS UMR 5292, Bron, Auvergne-Rhône-Alpes, France